CLINICAL TRIAL: NCT05181215
Title: A Single-Dose, Randomized, Open-Label, Two-Way Crossover, Bioequivalence Study of Bafiertam (Monomethyl Fumarate) 190 mg and Vumerity® (Diroximel Fumarate) 462 mg Delayed-Release Capsules in Fasting Healthy Male and Female Subjects
Brief Title: Bioequivalence Study of Bafiertam 190 mg and Vumerity® 462 mg Delayed-Release Capsules in Fasting Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Banner Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BLS-11-110
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — monomethyl fumarate; diroximel fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bafiertam (Experimental): 190 mg (2 x 95 mg) delayed-release capsules
  Interventions: Drug: Monomethyl Fumarate 190 Mg
- Vumerity (Active Comparator): 462 mg (2 x 231 mg) delayed-release capsules
  Interventions: Drug: Diroximel Fumarate 462 mg

INTERVENTIONS:
Drug: Monomethyl Fumarate 190 Mg — 2 x oral 95 mg capsules, delayed-release
  Other Names: Bafiertam®, BLS-11
  Arms: Bafiertam
Drug: Diroximel Fumarate 462 mg — 2 x 231 mg capsules, delayed-release
  Other Names: Vumerity®
  Arms: Vumerity

SUMMARY:
A single-dose, randomized, open-label, two-way crossover, two-period, two-sequence, two-treatment, single-center, bioequivalence study of Bafiertam and Vumerity.

DETAILED DESCRIPTION:
A single-dose, randomized, open-label, two-way crossover, two-period, two-sequence, two-treatment, single-center to assess the bioequivalence of Bafiertam (Monomethyl Fumarate) 190 mg (administered as 2 x 95 mg) Delayed-Release Capsules and Vumerity® (Diroximel Fumarate) 462 mg (Administered as 2 x 231 mg) Delayed-Release Capsules as assessed by plasma monomethyl fumarate concentrations in 40 healthy, non-smoking, male, and non-pregnant female volunteers under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking (at least for 6 months prior to first study drug administration) male and non-pregnant female volunteers, 18 years of age and older.
2. BMI that is within 18.5-33.0 kg/m², inclusive.
3. Healthy, according to the medical history, ECG, vital signs, laboratory results, and physical examination as determined by the PI/Sub-Investigator.
4. Systolic blood pressure between 95-140 mmHg, inclusive, and diastolic blood pressure between 55-90 mmHg, inclusive, and heart rate between 50- 100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
5. Clinical laboratory values within BPSUSA's most recent acceptable laboratory test range, and/or values are deemed by the PI/Sub-Investigator as "Not Clinically Significant".
6. Ability to comprehend and be informed of the nature of the study, as assessed by BPSUSA staff. Capable of giving written informed consent prior to receiving any study medication. Must be able to communicate effectively with clinic staff.
7. Ability to fast for at least 14 hours and consume standard meals.
8. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
9. Agree not to have a tattoo or body piercing until the end of the study.
10. Agree not to receive a vaccination (live attenuated vaccine) during the study and until 30 days after the study has ended (last study procedure).
11. Agree not to drive or operate heavy machinery if feeling dizzy or drowsy following study drug administration until full mental alertness is regained.
12. Female subjects must fulfill at least one of the following: Be surgically sterile for a minimum of 6 months; Post-menopausal for a minimum of 1 year; Agree to avoid pregnancy and use a medically acceptable method of contraception from at least 30 days prior to the study until 90 days after the study has ended (last study procedure).
13. Male subjects who are able to father children must agree to use medically acceptable methods of contraception during the study and for 90 days after his last study drug administration.

Exclusion Criteria:

1. Known history or presence of any clinically significant hepatic (e.g., hepatic impairment), renal/genitourinary (e.g., renal impairment), gastrointestinal, cardiovascular (supraventricular extrasystoles, atrioventricular block first degree, angina pectoris), cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.
2. Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first study drug administration, as determined by the PI/Sub-Investigator.
3. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the PI/Sub-Investigator.
4. Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
5. A positive test result for any of the following: HIV, Hepatitis B surface antigen, Hepatitis C, drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), alcohol test and cotinine. Positive pregnancy test for female subjects.
6. Known history or presence of: Alcohol or Drug abuse or dependence; Hypersensitivity or idiosyncratic reaction to monomethyl fumarate, diroximel fumarate, dimethyl fumarate, Bafiertam, Vumerity, their excipients, and/or related substances; Lymphocyte count <1.5x 10^9/L; Liver injury; Gastroenteritis; Protein in urine / Fanconi syndrome; Progressive multifocal leukoencephalopathy; Serious opportunistic infections, fungal infections; Food allergies and/or presence of any dietary restrictions unless deemed by the PI/Sub-I as "Not Clinically Significant"; Severe allergic reactions.
7. Intolerance to and/or difficulty with blood sampling through venipuncture.
8. Abnormal diet patterns (for any reason) during the four weeks preceding the study, including fasting, high protein diets, etc.
9. Individuals who have donated, in the days prior to first study drug administration: 50-499 mL of blood in the previous 30 days; 500 mL or more in the previous 56 days.
10. Donation of plasma by plasmapheresis within 7 days prior to first study drug administration.
11. Individuals who have participated in another clinical trial or who received an investigational drug within 30 days prior to first study drug administration.
12. Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing and containing grapefruit and/or pomelo within 10 days prior to first study drug administration.
13. Use of any prescription medication within 14 days prior to first study drug administration (except for hormonal contraceptives).
14. Use of antineoplastic, immunosuppressive, or immune-modulating therapies and fumaric acid derivatives, nephrotoxic drugs within 14 days prior to first study drug administration.
15. Use of any over-the-counter medications (including oral multivitamins, herbal, and/or dietary supplements) within 14 days prior to first study drug administration (except for spermicidal/barrier contraceptive products).
16. Individuals having undergone any major surgery within 6 months prior to the start of the study unless deemed otherwise by PI/Sub-Investigator.
17. Difficulty with swallowing the whole capsule.
18. Women who are pregnant or lactating.
19. Unable or unwilling to provide informed consent.
20. Have had a tattoo or body piercing within 30 days prior to first study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
The Bioequivalent (BE) Comparison of AUC0-inf of Monomethyl Fumarate (MMF) Between Treatments | 24 hours
  Pharmacokinetics: Plasma concentrations of MMF will be determined and used to calculate AUC0-inf MMF for each treatment. Venous blood samples were collected immediately prior to dosing (time 0), and then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 14, 16, 18, 20, 22, and 24 hours postdose.
The BE Comparison of Cmax of Monomethyl Fumarate (MMF) Between Treatments | 24 hours
  Pharmacokinetics: Plasma concentrations of MMF will be determined and used to calculate Cmax of MMF for each treatment. Venous blood samples were collected immediately prior to dosing (time 0), and then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 14, 16, 18, 20, 22, and 24 hours postdose.

CONTACTS AND LOCATIONS:
Overall Officials: Franck Rousseau, MD, Study Director — Banner Life Sciences LLC
Locations (1):
- BioPharma Services, Inc., St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No